CLINICAL TRIAL: NCT06454565
Title: Effects of Traditional Martial Arts, Open and Locked Exercise on the Physical and Mental Health of Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof., Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEE2024
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Drug Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Health Qigong - 12-Step Daoyin Health Preservation Exercises (Experimental): All classes are conducted offline and are implemented by professional Health Qigong instructors.
  Interventions: Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises
- Locked exercise (Experimental): All classes are held offline with professional instructors.
  Interventions: Behavioral: Locked exercise
- Multiplayer open exercise (Experimental): All classes are held offline with professional instructors.
  Interventions: Behavioral: Multiplayer open exercise
- Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with locked exercise (Experimental): All classes are held offline with professional instructors.
  Interventions: Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with locked exercise
- Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with open exercise (Experimental): All classes are held offline with professional instructors.
  Interventions: Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with open exercise
- Control group (No Intervention): Disseminating knowledge about the dangers of drugs

INTERVENTIONS:
Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises — All participants received a six-month intervention consisting of two phases: the first month was a movement learning and consolidation phase of 45 minutes per session, once a day; the second five months were a formal practice phase of 45 minutes per session, once a day. In the first phase, participants learn four new movements per session and consolidate these exercises in the next session. After learning all the movements, the remaining time of the first phase was used to consolidate the exercises. In the second phase, participants perform a full Health Qigong - 12-Step Daoyin Health Preservation Exercises practice in each session.
  Arms: Health Qigong - 12-Step Daoyin Health Preservation Exercises
Behavioral: Locked exercise — All participants received a six-month intervention of 45 minutes once a day. All participants performed blocked aerobic exercise.
  Arms: Locked exercise
Behavioral: Multiplayer open exercise — All participants received a six-month intervention in the form of a balloon game competition. The intervention consisted of two phases: the first month consisted of a movement learning and consolidation phase of 45 minutes per session, once a day; the second five months consisted of a formal competition phase of 45 minutes per session, once a day. In the first phase, coaches taught participants the technical movements and rules. In the second phase, participants competed in groups during each session, with the coaches acting as referees.
  Arms: Multiplayer open exercise
Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with locked exercise — All participants received the intervention for six months, 45 minutes each time, once a day. All participants performed blocked exercise followed by Health Qigong - 12-Step Daoyin Health Preservation Exercises. The schedule was consistent with the Health Qigong - 12-Step Daoyin Health Preservation Exercises group and the Blocked Exercise group.
  Arms: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with locked exercise
Behavioral: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with open exercise — All participants received the intervention for six months, 45 minutes each time, once a day. All participants performed multiplayer Open Exercise followed by Health Qigong - 12-Step Daoyin Health Preservation Exercises exercises. The schedule was consistent with the Health Qigong - 12-Step Daoyin Health Preservation Exercises group and the Multiplayer Open Exercise group.
  Arms: Health Qigong - 12-Step Daoyin Health Preservation Exercises combined with open exercise

SUMMARY:
The aim of this study is to discuss the efficacy of Chinese traditional martial arts in reducing drug addiction and improving the physical and mental health of drug addicts.

ELIGIBILITY:
Inclusion Criteria:

* Normal mental state, able to understand and accept instructions
* Drug users who have survived the detoxification period
* Without major diseases

Exclusion Criteria:

* Drug use for more than 2 years
* Drug abusers who have entered a drug rehabilitation center more than once

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Using a Jamar hydraulic hand dynamometer to investigate change of handgrip in participants. | Month 6
  Participants will receive a handgrip strength test before and after the intervention to assess the change from baseline handgrip strength at 6 months.
Using a step test to test participants' aerobic endurance. | Month 6
  Participants will undergo an aerobic endurance test before and after the intervention to assess the change in aerobic endurance from baseline at 6 months.
Using a spirometry tester to investigate changes in pulmonary capacity of the participants. | Month 6
  Participants will receive a spirometry test (vital capacity, ml) before and after the intervention to assess the change in spirometry from baseline at 6 months.
The participants' flexibility was tested by seated forward bending. | Month 6
  Participants will receive a seated forward bend test before and after the intervention to assess changes in flexibility from baseline at 6 months.
The participants reaction abilities were tested by means of a reaction time tester. | Month 6
  Participants will receive a response time test before and after the intervention to assess the change in responsiveness from baseline at 6 months.
The balance ability of the participants was tested through a one-legged standing test. | Month 6
  Participants will receive a one-legged standing test before and after the intervention to assess the change in balance from baseline at 6 months.
The core strength of the participants was tested through a sit-up test. | Month 6
  Participants will undergo a sit-up test before and after the intervention to assess changes in core strength from baseline at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China

REFERENCES:
- [Derived] Yang G, Meng D, He S, Wei M, Li M, Zhang L, Pan Z, Wang Z. Comparative effects of Health Qigong and closed motor exercise on the physical and mental health of female drug rehabilitation participants: a randomized controlled trial. BMC Complement Med Ther. 2025 Feb 4;25(1):38. doi: 10.1186/s12906-025-04797-y. PMID 39905407